CLINICAL TRIAL: NCT05893550
Title: Omega-3 Supplementation to Both Parent and Adolescent to Reduce Behavior Problems
Brief Title: Omega-3 Supplementation to Both Parent and Adolescent
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Joint Child Health Project, Mauritius (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JCHP-2
Record Dates: First submitted 2017-11-06; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Behavior Problems
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: 2 x 2 randomized, double-blind, stratified, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is double-blind. Neither the participant nor the caregiver not the outcomes Assessor will know which group the participant is assigned to. The local PI in Mauritius (Tashneem Mahoomed, National Director) will also be blind to treatment condition. Only the PI in Philadelphia will have knowledge of treatment assignment, and he has no contact with participants in Mauritius.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Both Parent and child (Experimental): Smartfish Omega Both parent and child receive Omega-3 drink
  Interventions: Dietary Supplement: Smartfish Omega
- Parent Only (Experimental): Smartfish Omega Only the parent receives Omega-3 drink, child receives Placebo.
  Interventions: Dietary Supplement: Smartfish Omega; Dietary Supplement: Smartfish Fruit Juice Only
- Child Only (Experimental): Smartfish Omega Only the child receives Omega-3 drink, the parent receives placebo
  Interventions: Dietary Supplement: Smartfish Omega; Dietary Supplement: Smartfish Fruit Juice Only
- Neither (Placebo Comparator): Smartfish Fruit Juice Only Neither parent nor child receives omega-3; both receive placebo (fruit juice).
  Interventions: Dietary Supplement: Smartfish Fruit Juice Only

INTERVENTIONS:
Dietary Supplement: Smartfish Omega — Fruit juice drink containing Omega-3: the experimental condition
  Arms: Both Parent and child; Child Only; Parent Only
Dietary Supplement: Smartfish Fruit Juice Only — this is a fruit juice drink with no omega-3 added. it is the placebo condition
  Arms: Child Only; Neither; Parent Only

SUMMARY:
The overarching, long-term goals are to develop a non-invasive biological approach to prevention of youth aggression, and ultimately adult violence.

The specific aims of this 2 x 2 randomized, double-blind, stratified, placebo-controlled trial of omega-3 supplementation to adolescents and caregivers are: (1) to investigate whether a nutritional intervention to adolescents and their parents can reduce externalizing behavior problems; (2) to examine the impact of a dual nutritional intervention to both parents and adolescents on adolescent externalizing behavior problems; (3) to identify mechanisms of action by which omega-3 supplementation impacts externalizing behavior in adolescents. It is expected that omega-3 supplementation will reduce adolescent behavior problems, and that dual supplementation to both the caregiver and adolescent will result in exponential improvements in adolescent behavior. A secondary prediction is that improvements in neurocognitive functioning will partially account for any behavioral improvements observed. Effects on scholastic ability are also explored.

DETAILED DESCRIPTION:
Despite increasing evidence for a significant neurobiological basis to aggression, biological interventions have been largely side-stepped, despite the fact that violence is a global public health problem. An important need is to develop socially acceptable ways of bettering brain functioning to reduce adolescent behavior problems, a critical developmental stage for adult violence perpetration and mental health problems. This is the primary health challenge that this proposal aims to tackle. Our pilot data documents that omega-3, a long-chain fatty acid which is critical for brain structure and function, reduces behavior problems in children and adolescents six months after the end of supplementation. If it can further document support and extension of the pilot findings with dual supplementation to both parent and adolescent, and if the investigators can begin to identify the mechanisms of action underlying change, this can provide a new vista on biological interventions for adolescent externalizing problems that predispose to violence. The overarching, long-term goals are to develop a non-invasive biological approach to prevention of youth aggression, and ultimately adult violence.

The specific aims of this 2 x 2 randomized, double-blind, stratified, placebo-controlled trial of omega-3 supplementation to adolescents and caregivers are: (1) to investigate whether a nutritional intervention to adolescents and their parents can reduce externalizing behavior problems; (2) to examine the impact of a dual nutritional intervention to both parents and adolescents on adolescent externalizing behavior problems; (3) to identify mechanisms of action by which omega-3 supplementation impacts externalizing behavior in adolescents. It is expected that omega-3 supplementation will reduce adolescent behavior problems, and that dual supplementation to both the caregiver and adolescent will result in exponential improvements in adolescent behavior. A secondary prediction is that improvements in neurocognitive functioning will partially account for any behavioral improvements observed. Effects on scholastic ability are also explored.

The paradigm-shift that could influence clinical practice is the use of a biological intervention that is not solely focused on the adolescent, but which is also applied to the primary caregiver. To the investigators' knowledge, such dual supplementation has never been examined. From an epidemiological standpoint, if this dual intervention approach could reduce even modestly the overall level of aggressive and antisocial behavior in the community at large, there is the promise of enhancing child health and development with a clinical paradigm novel in the biological study of behavior problems. The study's significance extends beyond adolescent behavior problems, which predispose not just to later adult violence, but also a wide array of adult psychiatric disorders. These adult outcomes result in an enormous societal burden in terms of economic costs, reduced occupational functioning, social functioning, and quality of life for both victims and perpetrators, a burden which could be significantly ameliorated if the pilot findings are supported.

ELIGIBILITY:
Inclusion Criteria:

* adolescents between Age 11 and 18
* willing to participate in a randomized control trial
* parent participated in prior Mauritius Child Health Project

Exclusion Criteria:

* Allergy to fish or fish products
* Intellectual disability
* Use of fish oil supplementations in the past 6 months

Ages: 11 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 800 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in behavior problems | 0, 6, 12, 18 months
  Behavior problems are assessed on a battery of measures with standardized units from parent and child reports. . Aggressive behavior, rule-breaking behavior, and attention problems will be assessed using the Youth Self-Report (YSR; Achenbach & Rescorla, 2001). The fourth scale is the 10-item version of the Inventory of Callous-Unemotional Traits (ICU; Ray et al., 2016). The final two scales are the Reactive and Proactive Aggression scales of the Reactive and Proactive Aggression Questionnaire (Raine et al. 2006). To reduce variables to a more reliable and all-encompassing construct of antisocial behavior, and to avoid Type 1 error, a principal components analysis was conducted on these six measures. Factor scores will be saved using the regression method, with higher scores indicating higher child antisocial behavior. Factor scores over time will be assessed.

SECONDARY OUTCOMES:
Change in neurocognitive functioning | 0,6,12,18 months
  assessed from a neuropsychological test battery: standardized units. The Digit Forward, Digit Backward, Coding, and Arithmetic, Pairing, and Free Recall tests will be administered using the Wechsler Intelligence Scale for Children (WISC-III; Wechsler, 1991), together with the Trails A and Trails B tests.Factor scores will be saved using the regression method, with higher scores indicating higher cold EFs. Chganges in factor scores over time will be evaluated.
Change in substance use. | 0, 6,12,18 months
  smoking, alcohol, marijuana: standardized units. These will be assessed based on the Achenbach Adult Self-Report. Change over time will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Raine, D.Phil., Principal Investigator — University of Pennsylvania; Tashneem Mahoomed, BSc, Study Director — Joint Child Health Project
Locations (1):
- Joint Child Health Project, Quatre Bornes, Mauritius

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Raine A, Liu J, Venables PH, Mednick SA, Dalais C. Cohort profile: The Mauritius Child Health Project. Int J Epidemiol. 2010 Dec;39(6):1441-51. doi: 10.1093/ije/dyp341. Epub 2009 Dec 7. No abstract available. PMID 19995862
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/19995862

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT05893550/Prot_SAP_000.pdf